CLINICAL TRIAL: NCT05830175
Title: The Effects Of Cervikal Mobilization On Balance And Gait Parameters In Individuals With Stroke
Brief Title: The Effects Of Cervical Mobilization
Acronym: CM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Erhan KIZMAZ, Msc. Phsyioterapist, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AZİZPAMUKKALE
Record Dates: First submitted 2023-03-20; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Stroke; Ischemic Stroke; Chronic Stroke
Keywords: cervical mobilization; head posture; gait parameters; balance; stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Demographic data, gait parameters, balance parameters and craniovertebral angle values of individuals were evaluated with clinical data evaluation form, Spatio-Temporal Gait Analysis (LEGSystm), Portable computerized kinesthetic balance device (SportKAT 550) and photometer, respectivelyThe evaluations were performed 2 times before and after the treatment.
  In addition to the 1 hour Bobath treatment, the study group received 15 minutes of cervical region joint and soft tissue mobilizations 3 times per week along 4 weeks. The control group was treated with Bobath 3 days per week along 4 weeks and each session was 75 minutes.
Who Masked: Participant
Masking Description: Basic randomization via SPSS v24.0 program
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Craniovertebral angle assesment (Experimental): Craniovertebral angle is the most widely used measurement to assess Forward head posture. Craniovertebral angle is described as the acute angle formed between a horizontal line passing through the spinous process of the seventh cervical vertebra (C7) and the line connecting the midpoint of the tragus to the spinous process of C7.
  Interventions: Other: manual therapy for cervikal region; Other: osteopathic suboccipital myofascial release technique
- Spatio-temporal gait analyz (LEGSystm) (Experimental): The gait performance of the cases was evaluated with a spatio-temporal gait analysis device named LEGSystm developed by BioSensicstm The device is controlled from the computer with its own software and instantly sends the raw data it collects to the computer via Bluetooth.The Modified Get Up and Go Test (MKYT), which is also supported by the legsyst, was used for assesment. The test was repeated 2 times and the average time was recorded. Legsystm provides information on double stride length, duration and speed of walking, as well as standing, turning, sitting times and total time.
  Interventions: Other: manual therapy for cervikal region; Other: osteopathic suboccipital myofascial release technique
- Portable computerized kinesthetic balance device (SportKAT 550) (Experimental): The gait performance of the cases was evaluated with a spatio-temporal gait analysis device named LEGSystm developed by BioSensicstm The device is controlled from the computer with its own software and instantly sends the raw data it collects to the computer via Bluetooth.The Modified Get Up and Go Test (MKYT), which is also supported by the legsyst, was used for assesment. The test was repeated 2 times and the average time was recorded. Legsystm provides information on double stride length, duration and speed of walking, as well as standing, turning, sitting times and total time.
  Interventions: Other: manual therapy for cervikal region; Other: osteopathic suboccipital myofascial release technique

INTERVENTIONS:
Other: manual therapy for cervikal region — Joint mobilization: In the stroke individuals included in the mobilization group, Grade 3 Central Posterior-Anterior (CPA) passive joint mobilization was applied with the Maitland method starting from the upper cervical region towards the lower cervical region, in 3 sets, 2 minutes and 1 minute rest.
  Other Names: mobilization of spine according to maitland concept
Other: osteopathic suboccipital myofascial release technique — The patient lies comfortably in the supine position. The therapist's forearms are supported on the treatment table, with the metacarpophalangeal and proximal interphalangeal joints flexed to approximately 45 degrees. After the therapist places his hands on the area where the patient's suboccipital muscles connect the occiput, he asks the patient to relax and rest his head on his fingers. Therapist pays attention to positioning the fingertips in suboccipital area No traction is performed during this technique. The position is maintained until the patient is relaxed. This treatment takes approximately 3-4 minutes.

SUMMARY:
The aim of this study is to examine the effects of cervical mobilization on balance and gait parameters in stroke individuals.

Twenty-four stroke individuals aged 30-65 years, with a mini mental test score of 24 and above, and with a maximum score of 3 according to the modified rankin scale, were included in this study. Individuals were randomly divided into 2 groups as study (Bobath approach and cervical mobilization n=12) and control group (Bobath approach n=12).

Demographic data, gait parameters, balance parameters and craniovertebral angle values of individuals were evaluated with clinical data evaluation form, Spatio-Temporal Gait Analysis (LEGSystm), Portable computerized kinesthetic balance device (SportKAT 550) and photometer, respectivelyThe evaluations were performed 2 times before and after the treatment.

DETAILED DESCRIPTION:
The aim of this study is to examine the effects of cervical mobilization on balance and gait parameters in stroke individuals.

Twenty-four stroke individuals aged 30-65 years, with a mini mental test score of 24 and above, and with a maximum score of 3 according to the modified rankin scale, were included in this study. Individuals were randomly divided into 2 groups as study (Bobath approach and cervical mobilization n=12) and control group (Bobath approach n=12).

Demographic data, gait parameters, balance parameters and craniovertebral angle values of individuals were evaluated with clinical data evaluation form, Spatio-Temporal Gait Analysis (LEGSystm), Portable computerized kinesthetic balance device (SportKAT 550) and photometer, respectivelyThe evaluations were performed 2 times before and after the treatment.

In addition to the 1 hour Bobath treatment, the study group received 15 minutes of cervical region joint and soft tissue mobilizations 3 times per week along 4 weeks. The control group was treated with Bobath 3 days per week along 4 weeks and each session was 75 minutes.

ELIGIBILITY:
Inclusion Criteria:

Individuals diagnosed with stroke beetwen 30-70 ages had hemiparetik lezion

Exclusion Criteria:

Having previously diagnosed orthopedic diseases related to the spine

* Acute or chronic infections (including HIV)
* Serious pathologies (such as cancer, spondylolisthesis, rheumatoid arthritis or ankylosing spondylitis)
* Have a history of whiplash or cervical surgery
* Having diseases that cause balance weakness (spinal cord damage, cerebellar ataxia, Parkinson's disease)
* Having another neurological disease
* Having a vision problem
* Receiving another treatment that will affect balance and walking
* Having a vision problem
* Receiving another treatment that will affect balance and walking

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-03-15 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
forward head posture | during the procedure
  Craniovertebral angle assesment Craniovertebral angle is the most widely used measurement to assess Forward head posture. Craniovertebral angle is described as the acute angle formed between a horizontal line passing through the spinous process of the seventh cervical vertebra (C7) and the line connecting the midpoint of the tragus to the spinous process of C7.
gait parameters analyz | during the procedure
  We evaluated the gait performance of the subjects using the spatio-temporal gait analysis device called LEGSystm developed by BioSensics. The device consists of two sensors that are placed with Velcro about 3-5 cm above the subject's ankle. The device is controlled from a computer through its software, and the raw data it collects is sent to the computer via Bluetooth in real-time. The software analyzes the raw data collected by the device and converts it into results. For evaluation, we used the Modified Get Up and Go Test , which is supported by the device. We recorded the average times of the test by repeating it twice. LEGSystm provides information on the length, duration, and speed of walking, as well as the time for standing up, turning, sitting, and the total time .
balance assesment | during the procedure
  SporKAT examines the balance in 2 main parameters as static and dynamic, and 4 main parameters as forward-backward, right-left. SporKAT consists of a platform on the ground and a screen designed to face the patient, 1 meter away from the patient. Before the individual to be evaluated is taken to the platform, the pressure of the platform is adjusted, the increase in the pressure value stabilizes the platform and reduces its ability to disrupt the balance parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Aziz Dengiz, Denizli, Pamukkale, Turkey (Türkiye)